CLINICAL TRIAL: NCT03504046
Title: Inpatient Safety and Feasibility Evaluation of the Zone-MPC Control Algorithm Integrated Into the APS APP
Brief Title: Safety and Feasibility Evaluation of the APS APP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G180011
Record Dates: First submitted 2018-04-05; First posted 2018-04-20 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: artificial pancreas; hyperglycemia; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Artificial Pancreas App (Experimental): After completing a 1 week open-loop run in period, subjects will use the APS APP for a 48-hour period in an observed transitional environment.
  Interventions: Device: Artificial Pancreas App

INTERVENTIONS:
Device: Artificial Pancreas App — The portable Artificial Pancreas System App (APS APP) is an artificial pancreas system comprised primarily of an insulin pump, a continuous glucose monitor (CGM), and a cellular phone device to connect the components.

SUMMARY:
This clinical trial is a safety and feasibility study to assess the performance of artificial pancreas (AP) system using the Zone Model Predictive control (Zone-MPC) and Health Monitoring System (HMS) algorithms embedded into the APS APP platform.

DETAILED DESCRIPTION:
The system will be evaluated on up to 10 adult subjects with type 1 diabetes age 18-75 years old at a single clinical site (Sansum Diabetes Research Institute), who will complete a 48-hour closed-loop (CL) session in an observed CRC environment with medical staff present. During the session subjects will bolus for all meals and snacks and perform a 45-minute walking session while supervised by medical staff. The AP system used consists of an insulin pump, a CGM sensor, and a phone app (the Artificial Pancreas System [APS] phone app).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years at the time of screening.
* Clinical diagnosis of type 1 diabetes for at least one year.
* Has been using an insulin pump for at least 6 months at the time of screening.
* HbA1c < 10.5%.
* Bolus for all meals and snacks that contain ≥ 5 grams of carbohydrate.
* Willing to perform at least 7 fingerstick blood glucose tests a day.
* If using Apidra (insulin glulisine) at home and planning to use the Tandem t:AP pump for the closed-loop session, willing to switch to Novolog or Humalog for the closed-loop session.
* Willing to refrain from taking acetaminophen products for the duration of the clinical trial.
* Willing to abide by the study protocol and use study-provided devices, including the Omnipod OR Tandem Pump, Dexcom CGM, glucometer, ketone meter and APS APP on the study phone device.

Exclusion Criteria:

* Pregnancy
* One or more episodes of hypoglycemia requiring an emergency room visit or hospitalization in the past 6 months.
* One or more episodes of hyperglycemia requiring an emergency room visit or hospitalization in the past 6 months.
* Known unstable cardiac disease or untreated cardiac disease, as revealed by history or physical examination.
* Dermatological conditions that would preclude wearing a CGM sensor or Pod/infusion site.
* One or more seizures in the past year.
* Any condition that could interfere with participating in the trial, based on investigator judgment.
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Percent time in glucose range 70-180 mg/dL | 48 hours
  Time in target glucose range overall

SECONDARY OUTCOMES:
Percent time in glucose range 80-140 mg/dL overnight | 48 hours
  Overnight time in tight target range
Percent time in glucose range 70-150 mg/dl postprandial within 5 hours following meals | 48 hours
  Post prandial time in target
Percent time glucose < 70 mg/dL | 48 hours
  Hypoglycemia
Percent time glucose < 54 mg/dL | 48 hours
  Significant Hypoglycemia
Percent time glucose > 180 mg/dL | 48 hours
  Hyperglycemia
Percent time glucose > 250 mg/dL | 48 Hours
  Significant Hyperglycemia
Connectivity Analysis (Number of Connection Errors Between devices) | 48 Hours
  Failure analysis of the devices/connectivity issues that may occur. This includes the overall number of connectivity errors between pump, sensor and phone device and the types of errors and how they were addressed.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Dassau, PhD, Principal Investigator — Harvard University; Jordan Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No